CLINICAL TRIAL: NCT02349932
Title: The Influence of Histo-blood Group Antigen Polymorphism on the Composition of the Microbiota
Status: Withdrawn | Type: Observational
Why Stopped: Expired with IRB (2/2/2019).
Sponsor: University of Florida (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201400446-N; R01AI116892 (NIH)
Record Dates: First submitted 2015-01-23; First posted 2015-01-29 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Microbiota Analysis in Healthy Subjects

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, saliva, and fecal material will be collected from subjects. The blood and saliva will be used for typing sugar expression. DNA will be extracted from stool samples and used for characterization of the gut flora.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Adults: The following samples will be collected: fecal, blood, and saliva
  Interventions: Other: Healthy Adults

INTERVENTIONS:
Other: Healthy Adults — The following samples will be collected: fecal, blood, and saliva. The samples will be tested for HBGA-reactive antigens using an immunoaffinity assay.

SUMMARY:
A person's blood type is defined by the types of sugars they express on their red blood cells, with antibodies being made to non-self sugars and excluding blood cells expressing these sugars (the basis of blood transfusion reactions). These same sugars can be expressed by commensal bacteria in our gut lumens. The investigators hypothesize that a person's antibodies to non-self sugars also attach to and exclude non-self sugar-expressing bacteria in our guts. Supporting our hypothesis, a person's blood type correlates with the overall composition of their gut flora. Because these sugars are also used by certain pathogens to initiate infection, this information could directly inform our understanding of host susceptibility to various infectious organisms.

DETAILED DESCRIPTION:
A member of the study staff will collect a small volume of blood sample through a finger prick and 2-3 milliliters of saliva from you. Using these samples, we will determine your blood type (defined by your expression of specific sugars on your red blood cells) and your expression pattern of these sugars in body secretions (e.g., saliva). You will provide us with a fecal sample collected the day of your appointment. The fecal sample should be collected in a pre-provided collection container and should be collected within 12 hours of drop-off. Using your fecal sample, we will determine the types of bacteria present in your normal gut flora and whether they express the same sugars expressed on your blood cells. Tests will be done only for research purposes and will not be evaluated or used to diagnose or treat any of your medical problems. Sample collection may need to be repeated if required for your medical care in the future.

ELIGIBILITY:
Inclusion Criteria:

* healthy,
* adult

Exclusion Criteria:

* younger than 18,
* older than 60,
* pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Blood typing (Blood and saliva will be used to determine overall blood type) | 1 day
  Blood and saliva will be used to determine overall blood type.
Quantitative PCR (PCR will be used to enumerate commensal bacteria in fecal samples) | 1 day
  PCR will be used to enumerate commensal bacteria in fecal samples

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie M Karst, Ph.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States